CLINICAL TRIAL: NCT01541644
Title: A Pilot Study to Evaluate the Efficacy and Explore the Mechanism of Acupuncture in Treating Bortezomib-induced Peripheral Neuropathy (BIPN) in Multiple Myeloma Patients
Brief Title: 1068GCC Evaluate Efficacy & Explore Mechanism of Acupuncture in Treating Bortezomib-induced Peripheral Neuropathy (BIPN) in Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00047788; GCC 1068 (Other: University of Maryland Greenebaum Cancer Center)
Record Dates: First submitted 2012-02-20; First posted 2012-03-01 (Estimated); Results first posted 2016-03-11 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Peripheral Neuropathies; Multiple Myeloma
Keywords: Acupuncture Therapy; bortezomib-induced peripheral neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases; Multiple Myeloma | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Acupuncture (Experimental): All participants will receive acupuncture treatments over a total of 10 weeks.
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — Participants will receive acupuncture treatment twice weekly for 2 weeks, then once per week for 4 weeks, and then biweekly for 4 weeks.

SUMMARY:
Patients are asked to be in this study if they have multiple myeloma and are having tingling, numbness and pain from taking bortezomib (velcade®). Patients who have been diagnosed with multiple myeloma often take bortezomib (velcade®).

This research is being done to find out if acupuncture can reduce the nerve pain, tingling, and/or numbness patients experience due to bortezomib (velcade®).

Acupuncture is a medical technique of inserting very thin needles into the "energy points" on the body with the aim to restore health and well-being. It has been used widely to treat pain, such as lower back pain and nerve pain. In this study we will see if acupuncture can be used to ease nerve pain and tingling, numbness that is caused by bortezomib.

DETAILED DESCRIPTION:
Information gained from this clinical trial will provide insight into the efficacy and mechanism of acupuncture in reducing Bortezomib-induced Peripheral Neuropathy (BIPN) in multiple myeloma patients. It will examine the effect of acupuncture on serum proinflammatory cytokine and β-endorphin levels to further understand the mechanism of acupuncture on a molecular level. This study is the first clinical trial studying the effect of acupuncture on treating BIPN. It is also the first study to explore the mechanism of acupuncture through frequent small amount of blood draws at six time points to detect changes in proinflammatory cytokines and β-endorphins. It has the potential to identify a minimal risk non-pharmacological intervention to alleviate BIPN symptoms, and to significantly improve our understanding of the mechanism of acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of multiple myeloma.
* Greater than or equal to grade 2 BIPN as defined by the National Cancer Institute - -Common Toxicity Criteria (NCI-CTC) 4.0.
* BIPN symptoms persist after bortezomib has been discontinued.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-3.
* Men and women who are ≥ 18 years old
* The patient is aware of the nature of his or her diagnosis, understands the study regimen, its requirements, risks, and discomforts, and is able and willing to sign an informed consent form.

Exclusion Criteria:

* Prior acupuncture within the past month.
* Life expectancy is < 3 months.
* Plan to go on experimental drug for multiple myeloma that is known to cause peripheral neuropathy in the next 14 weeks.
* Concomitant treatment with chemotherapy, unless approval is given by the Principal Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ting Bao, MD, DABMA, Principal Investigator — University of Maryland Marlene & Stewart Greenebaum Cancer Center
Locations (1):
- University of Maryland Marlene & Stewart Greenebaum Cancer Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acupuncture
Started | 27
Completed | 24
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Acupuncture
Number analyzed (Participants) | 27
Age, Customized [Mean (Full Range); unit: years] | 63 [49 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Response Rate (Via FACT/GOG-Ntx Scores) Effectiveness and Safety of Acupuncture in Alleviating Neuropathic Symptoms When Treating Patients With Moderate to Severe Bortezomib-induced Peripheral Neuropathy (BIPN)
Description: The Neuropathic Pain Scale (NPS) uses self-report visual analogue scales (VAS) to quantify on a scale of 0-10 (with total NPS score of 1-100), global pain intensity and unpleasantness and 8 other descriptive qualities of neuropathic pain. Response defined as average change of Clinical Total Neuropathy Score (TNSc) greater than or equal to 10% over 10 weeks compared to baseline. Effect defined as as average change of Functional Assessment of Cancer Therapy-Neurotoxicity/ Gynecologic Oncology Group (FACT/GOG-Ntx)over 10 weeks as compared to baseline. Safety will be assessed by recording side effects from acupuncture treatment. Please note TNSc results deemed invalid as original validation of TNSc was performed by 2 neuromuscular trained physicians & the TNSc in our trial was performed by a research nurse. The reliability & validity of research nurse's TNSc not established pre-trial. For the scale range, the higher the score the worse the symptoms and function. No subscales were used.
Time Frame: Baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale (1 - 100)
Arm/Group | Acupuncture
Number analyzed (Participants) | 27
units on a scale (1 - 100) | 13.3 (6.5)

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Acupuncture
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

LIMITATIONS AND CAVEATS:
TNSc results deemed invalid as original validation of TNSc was performed by 2 neuromuscular trained physicians & the TNSc in our trial was performed by a research nurse. The reliability & validity of research nurse's TNSc not established pre-trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes